## Informed Consent Form of the First Affiliated Hospital of Zhengzhou University

Efficacy of sequential donor infusion of lymphocyte therapy in patients research topic relapsed after allogeneic hematopoietic stem cell transplantation for acute B lymphocytic leukemia Ward 5, Hematology Department, Haemopoietic Stem Cell Transplant The applicant Center, the First Affiliated Hospital of Zhengzhou University (1) C RO Scheme number v 1.1 Scheme version number V 1.1 on November 15,2023 and version date The name of the research The First Affiliated Hospital of Zhengzhou University institution Research institution 43 University Road, Zhengzhou city, Henan Province address Principal investigator Bian Zhilei contact number 0371-668622 Patient name abbreviation Patient Screening Number

### Instructions for the subjects

#### Dear subject:

You will be invited to attend a by the first affiliated hospital of Zhengzhou university hematopoietic stem cell transplantation center hematology five ward (1), the center hosted by PI of clinical research, is to prove that belin or sequential donor lymphocyte infusion therapy in acute B lymphocyte leukemia allogeneic hematopoietic stem cell transplantation relapse in patients with curative effect of a study. Scientific Research and Clinical Trials Ethics Committee of the First Affiliated Hospital of Zhengzhou University Address: No.43, University Road, Zhengzhou City, Henan Province Tel: 0371-66295219

Page number (page 1 of 6)18

Please read the following information carefully and, if you feel necessary, consult with your friends and family about your participation in this clinical study. Once all your questions are answered, you are satisfied with the explanation of the study and you decide to participate, you will need to sign this informed consent form. Participation in the clinical study is your voluntary activity, and you may agree to participate or disagree, and you may voluntarily withdraw from the clinical study at any time. The study was approved by the Ethics Committee of the First Affiliated Hospital of Zhengzhou University for the clinical study.

#### 2. Study objectives:

Acute lymphoblastic leukemia (ALL) is a malignant hematological disorder

Chemotherapy as well as hematopoietic stem cell transplantation. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the effective or even the only means to cure ALL and other malignant hematological diseases, but it still has a high recurrence rate after allogeneic acute lymphoblastic leukemia hematopoietic stem cell transplantation, and the prognosis of relapsed patients after transplantation is very poor, with an average survival time of about 5.5 months. There is no uniform treatment plan for relapsed patients after allogeneic HSCT. Donor lymphocyte infusion (DLI) is the primary salvage therapy for post-transplant relapse, but in the treatment of ALL patients, less than 20% of patients achieve reremission. Recurrence after ALL allogeneic HSCT is still an urgent clinical problem.

Belintouzumab is the first CD19 positive and CD3 positive targeted immunotherapy drug approved by the US FDA, and has also been approved for relapsed or refractory B-ALL in adults and children in China. By connecting CD3 on the T cell receptor complex with CD19 expressed on B cell line-derived cells, belintoeuromab clusters T cells with target

cells by forming cytolytic synapses, thereby activating endogenous T cells and enabling them to directional resolve CD19 + cells to achieve tumor cell killing. Belintuzumab in an effective salvage therapy for refractory acute B lymphoblastic leukemia in this patient population.

In this study, sequential DLI after acute B lymphoblastic leukemia allogeneic hematopoietic stem cell transplantation relapse (including MRD relapse and hematology relapse), observe the overall survival, disease-free survival, complications, adverse reactions and other indicators, explore the treatment plan of patients with acute B lymphoblastic leukemia allogeneic hematopoietic stem cell transplantation relapse.

#### 3. Study process and methods:

Acute B lymphocytic leukemia (B-ALL), seen regularly after allogeneic hematopoietic stem cell transplantation, was treated with sequential donor lymphocyte infusion (DLI).

For patients with positive MRD, belintouzumab 28  $\,\mu$  g 5-15 days was followed by DLI (MNC infusion was approximately 510 ^ 7 / kg to 110 ^ 8 / kg).

In patients with hematologic relapse, belintoeuromab 9  $\mu$  g d1-4,11.66  $\mu$  gd 5-7,28  $\mu$  gd 8 (8 to 21 days) before DLI (MNC infusion was approximately 510 ^ 7 / kg to 110 ^ 8 / kg).

#### 4. Potential benefits of the study:

Acute B lymphocytic leukemia (B-ALL) allogeneic hematopoietic stem cell transplantation has a very poor prognosis and a short survival. After treatment with this clinical study, your disease may be alleviated, causing prolonged survival, but it may not be effective. We cannot guarantee that can improve your health, but you participate in the study data, will be acute B lymphocyte leukocyte patients after heterogenic hematopoietic stem cell transplantation relapse treatment options to

provide evidence, in the future may help people who need treatment, increase the understanding of human physiology and behavior and benefit the whole society.

#### 5. Study risks and discomforts:

You may feel uncomfortable or risky during certain examinations, such as:

- 1. Collect blood samples: drawing blood from the arm may cause pain, swelling, slight dizziness and rare infection.
- 2. Bone marrow puncture: the site of bone marrow collection may cause pain and infection of the puncture site.

About the study drug:

Side effects can occur when using any drug. Your study doctor will ask if you have any side effects during each treatment. The risks of this clinical study are adverse effects of treatment with belintuzumab and DLI. Based on the information observed in previous clinical trials, it is speculated that the following adverse reactions may occur during the clinical studies, which may vary from person to person. Your study doctor may recommend that you suspend the study drug and treat you accordingly to control your adverse effects.

- (—) Belintoeuzumab related adverse reactions (detailed see belumab instructions) 1. cytokine release syndrome 2. nervous system toxicity 3. infection 4. tumor lysis syndrome 5. neutropenia and febrile neutropenia 6. The impact on driving and use of mechanical ability 7. The liver enzymes rise 8. pancreatitis 9. leukoencephalopathy, etc.
- (二) DLI adverse effects: myelosuppression, graft versus-host disease, infection, etc.

In addition, there may be currently unknown adverse reactions or risks. You will be promptly informed of any important new information that may affect your willingness to continue in this study.

#### 6. Other alternative treatment methods:

You can choose not to participate in this study, you can choose traditional chemotherapy or accept other clinical trials.

#### 7. Privacy protection:

If you decide to participate in this study, the study doctor and other investigators will use your medical information. This information may include your name, address, telephone number, medical history, and information obtained at your study follow-up. In the study analysis process and the published study results, your name and other information with relevant identity identification records will be kept confidential and not publicly used. Information that can identify you will not be disclosed to members outside of the study team without your permission. To ensure that the study is conducted as required, members of the Ethics Review Committee may access your personal data at the study site if necessary.

#### 8. Expenses and compensation:

In the course of your participation in the study, the expected risks arising in this study are all common complications of conventional treatment after allogeneic HSCT or after allogeneic HSCT. This study is an observational study that does not increase invasive procedures in subjects while not increasing patient treatment risk. So there is no additional compensation for this clinical study.

#### 9. Free to exit:

As a subject, you may be informed of the information and progress of the study and voluntarily decide to (continue) or not (continue). After participation, regardless of whether the injury occurred or was serious, you may choose to notify the investigator to withdraw from the study. The data after your withdrawal from the study will not be included in the study results, and any medical treatment and interests will not be affected. If you continue to participate in the study, the investigator will also discontinue the study.

If you have questions about the study content, please contact the study doctor at \_\_0371-66862272\_\_\_\_\_; if you have questions related to your rights, contact the ethics committee at the footer of the informed consent form.

# Informed Consent Form of the First Affiliated Hospital of Zhengzhou University

I have carefully read the informed consent form for the "efficacy of sequential donor lymphocyte infusion therapy in patients who relapse after allogeneic hematopoietic stem cell transplantation". I have had the opportunity to ask and all questions have been answered. I understand that participation in this trial is voluntary, I may choose not to participate in this trial or withdraw at any time after notifying the investigator without discrimination or retaliation, and any of my medical treatment and interests will not be affected. If I need any other diagnosis / treatment, or if I fail to comply with the trial plan, or for other reasonable reasons, the investigator may terminate my continued participation in this clinical trial. I voluntarily agree to participate in this clinical trial, and I will receive a signed copy of the "informed consent form".

Please copy: "I have read and understood this clinical trial and have volunteered for this clinical trial".

| Subject Name (block | |
|---|---|
| letters): | |
| Subjects signed: | |
| Subject ID Number: | |
| contact number: | |
| date: | yearmoonsun |
| (When the subject has insufficient or inst | ufficient informed consent ability, add |
| Name of guardian (kai kai): | |
| Signature of guardian: | |
| Guardian ID Number: | |

| Informed Consent Form Version Number: v 1.0 Date of the First Affiliated Hospital of Zhengzhou University: November 15,2023 | |
|---|---|
| Relationship with the | |
| subjects: | |
| contact number: | |
| date: | yearmoonsun |
| (When the subject or his guardian is not | reading, add or replace the following:) |
| Name of the Fair Witness (in | |
| regular letters): | |
| Signature of the Fair | |
| Witness: | |
| Fair Witness ID Number: | |
| contact number: | |
| date: | yearmoonsun |
| I have accurately informed the subject of the informed consent form and answered | |
| the questions, and the subject voluntarily participated in this clinical trial. And | |
| gave him a copy of the signed informed consent form. | |
| Study doctor Name (block | |
| letters): | |
| Signature of the study | |

\_\_\_\_year\_\_\_moon\_\_\_sun

physician:

date:

contact number: